CLINICAL TRIAL: NCT04139408
Title: A Prospective, Multicenter, Single Group Clinical Study to Evaluate the Safety and Effectiveness of Disposable Pulmonary Surgical Markers in the Localization of Pulmonary Nodules
Brief Title: Safety and Effectiveness of Disposable Pulmonary Surgical Markers in the Localization of Pulmonary Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Broncus Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-HM-01
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer
Keywords: Pulmonary Nodule; Localization; Marker
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disposable Pulmonary Surgical Marker (Experimental): Locate the pulmonary nodules with Disposable Pulmonary Surgical Marker before VATS.
  Interventions: Device: Disposable Pulmonary Surgical Marker

INTERVENTIONS:
Device: Disposable Pulmonary Surgical Marker — The subjects will undergo Marker placement procedure, within 24h before VATS.

SUMMARY:
During the VATS procedure, some pulmonary nodules are relatively small or far away from the pleura, resulting that they are difficult to be accurately located during the procedure.

The aim of this study is to evaluate the efficacy and safety of using disposable pulmonary surgical markers to localize pulmonary nodules in subjects prior to the resection of pulmonary nodules by video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
It is a prospective, multicenter, single group target value clinical trial. The subjects will undergo VATS within 24h after the placement of the Marker, then the Marker and targeted nodule will be removed during VATS. Subjects will be followed up intraoperatively, immediately after placement procedure to the end of VATS resection, 7 days after placement procedure/before discharge (whichever occurs earlier), and 30 days after Marker placement procedure. Demographic and baseline information of subjects, immediate operation success rate of marker placement, positioning success rate, and adverse events will be collected and recorded in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old；
* Pulmonary nodule, which satisfying any of the following Criteria:

  * solid nodules with diameter ≤1 cm or solid component ≤1 cm non-purely ground glass, and the distance between the solid component of the nodule and the visceral pleural>0.5cm;
  * Pure ground glass opacity (pGGO)；
  * Before VATS operation, the doctor judge that the nodule is difficult to locate during the operation.
* Pulmonary wedge resection or Segmental pulmonary resection under VATS is proposed;
* Preoperative evaluation shows that placing marker through bronchus is feasible；
* The subject is able to fully understand the requirements of clinical research;
* Subject or the legal representative signs the informed consent form.

Exclusion Criteria:

* Contraindications for bronchoscopy;
* Systemic factors: sepsis, history of repeated pulmonary infections, and any type of severe infectious disease within one month of screening；
* Severe cardio and pulmonary disease；
* Coagulation dysfunction, with a clear tendency to bleed;
* General anesthesia contraindication;
* Allergic history of nickel-titanium materials;
* Breast-feeding or may be or plan to be pregnant during the trial;
* Participating in clinical trials of other drugs or medical devices;
* Other conditions that Investigator consider the subject to be inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Positioning success rate | Immediately after VATS
  The proportion of patients who complete VATS resection of target pulmonary nodules/number of patients receiving localization of target pulmonary nodules before operation, expressed as "rate", will be evaluated during and immediately after surgery to evaluate the effectiveness of disposable pulmonary surgical markers in the localization of pulmonary nodules in surgery.

SECONDARY OUTCOMES:
Positioning success rate (in terms of marker placement) | Immediately after VATS
  The proportion of target pulmonary nodules underwent VATS resection/number of pulmonary nodules receiving localization before operation, expressed as "rate".
Immediate operation success rate of marker placement (in terms of marker, placement),including the following operations: | Immediately after marker placement
  1. The marker conveyor goes through the bronchoscope and reaches the target release position
  2. Marker is successfully released
  3. Fully retract the conveyor
  Complete all the above steps and record the success of the operation as "rate".
Operation time of Marker placement (in terms of marker placement) | Immediately after marker placement
  Defined as starting from the time the marker conveyor is inserted into the bronchoscope until it is withdrew from the bronchoscope.
Operation time of marker release through bronchoscopy (in terms of marker placement) | Immediately after marker placement
  Defined as starting from the time when the bronchoscope is inserted into the airway to the time when the marker conveyor is removed from the bronchoscope.
Operation time of exploration and removal of target lesion during VATS (in terms of marker placement) | Immediately after VATS
  Defined as starting lesion location exploration after the completion of preoperative surgical preparation and VATS access ports made, to the time of resection and removal of lung tissue.
Safety: AEs (Adverse Events) and SAEs (Serious Adverse Events) occured during the clinical trial | 30days
  AEs and SAEs occured from marker placement to 30days after the placement procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Qiu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Yunnan Cancer Hospital, Kunming
  - Cancer Hospital of Chinese Academy of Medical Sciences,Shenzhen Center, Shenzhen

IPD SHARING:
Plan to Share IPD: No